CLINICAL TRIAL: NCT05616026
Title: Short-messaging Services (SMS) Text for Uncontrolled Diabetes Among Persons Experiencing Homelessness
Brief Title: Texts for Diabetes Control Among Homeless Persons
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Ramin Asgary, Associate Professor School oh Public Health, PI, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: #11-21-ICTSHD-16
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Homelessness; SMS text; mobile Health; Clinical trial; Health disparities
MeSH Terms: conditions — Diabetes Mellitus | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Intervention versus Control group; Randomized at the Individual level
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention (INT) will include 6 months of DM management support via SMS texts including reminders for medication adherence, appointments, and DM self-care activities as well as education, and support.
  Interventions: Behavioral: Intervention
- Control (Placebo Comparator): The control (CL) will receive 6 months of texts for general health promotion.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Intervention — 6 months of diabetes management support via SMS texts including reminders for medication adherence, appointments, and diabetes self-care activities as well as education, and support
  Other Names: Diabetes SMS text
  Arms: Intervention
Behavioral: Attention Control — 6 months of texts for general health promotion
  Arms: Control

SUMMARY:
This mixed method study includes a Randomized Controlled Trial (RCT) and qualitative methods to assess the impact of a SMS text strategy in diabetes control among persons who experience homelessness.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is common among persons experiencing homelessness (PEH), often inadequately managed, and carries significant costs. SMS strategies for DM have not been tested among PEH despite the accessibility of mobile phones. This study uses a SMS strategy to offer better communication, education, and information management; improve outreach; facilitate care coordination; explore barriers to care; and support behavior changes. This mixed-methods (RCT and qualitative) study will be implemented in shelter-clinics in New York City in collaboration with community organizations, allowing for sustainability and scalability. Aim 1 will evaluate the efficacy of a 6-month SMS program for DM management versus an attention control on changes in HbA1c and adherence to DM self-care activities, medications, and appointments at 9 months in adult PEH with uncontrolled DM (n=100). Outcomes will be measured at 0, 3, 6, &9 months. Aim 2 will assess patients' and providers' attitudes, acceptability, and experience of the program through semi-structured interviews with PEH and providers.

ELIGIBILITY:
Inclusion Criteria:

* Homeless person age ≥ 21
* Diagnosed with type 2 DM
* Most recent visit HbA1c ≥ 8%
* English/Spanish speaking
* Connected to study sites' shelter-clinics for care

Exclusion Criteria:

* Pregnant or within 3 months postpartum
* Has an uncontrolled severe illness
* Has had a heart attack or stroke in the previous 6 months
* Inability to read/respond to texts
* Inability to provide informed consent
* Receiving inpatient care for severe substance abuse

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 9 months
  Hemoglobin A1c level

SECONDARY OUTCOMES:
Proportion of Days Covered (PDC) | 9 months
  Medication Adherence through Proportion of Days Covered of Medications
Appointment Adherence | 9 months
  Proportion of appointment adherence

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - George Washington University, Washington D.C., District of Columbia
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: No